CLINICAL TRIAL: NCT02955875
Title: Impact of Pharmaceutical Care Service for Type 2 Diabetes Mellitus Patients in Korea
Brief Title: Pharmaceutical Care Service in Diabetes
Acronym: IMPACT4-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hyun Yoon, Associate professor, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PNU-2014-001
Record Dates: First submitted 2016-10-26; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Pharmaceutical Services
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Pharmaceutical care (Experimental): Participants received systematically organized pharmaceutical care services, which were provided by pharmacists, in addition to the usual care. The usual care includes traditional consultation with pharmacists as well as traditional medical services provided by physicians, nurses, and dietitian.
  Interventions: Behavioral: Pharmaceutical care
- Usual care (No Intervention): Participants received the usual care, which includes traditional consultation with pharmacists as well as traditional medical services provided by physicians, nurses, and dietitian.

INTERVENTIONS:
Behavioral: Pharmaceutical care — Outpatient drug history management, drug regimen review, patient counseling and education before and/or after physician evaluation on the day of facility visit
  Other Names: Pharmaceutical service
  Arms: Pharmaceutical care

SUMMARY:
The purpose of this study is to examine the effectiveness of pharmaceutical care service in the management of poorly controlled type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria: Patients who visit Endocrinology and Metabolism department of Pusan National University Hospital, are with type 2 diabetes mellitus, and meet one of the following criteria

* Who are diagnosed with type 2 diabetes mellitus for the first time
* Who need the education for medication or disease
* Who are with poorly controlled blood glucose
* Who have poor medication adherence
* Who have been hospitalized with diabetes complication or poorly controlled blood glucose
* Whose physician recommend the pharmaceutical care to them

Exclusion Criteria: Patients who meet one of the following criteria

* Who are with gestational diabetes
* Who are not able to respond to questionnaires
* Who are with severe condition such as cerebrovascular disease, mental disorder, and acquired immune deficiency syndrome
* Who are not able to be followed-up during 9 months in Pusan National University Hospital

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Medications knowledge at 9 months | 9 months
  Patients' knowledge about diabetes medications was measured by an instrument. The instrument includes items such as the name of medication, mechanism of action, dosage, and side effects.

SECONDARY OUTCOMES:
HbA1c level at 9 months | 9 months
Random blood glucose level at 9 months | 9 months
Blood pressure at 9 months | 9 months
Cholesterol level at 9 months | 9 months
Proportion of participants taking statins 9 months | 9 months
Proportion of participants managing diabetes complications at 9 months | 9 months
Morisky Medication Adherence Scale at 9 months | 9 months
5-level version of the EQ-5D at 9 months | 9 months
EQ Visual Analogue Scale at 9 months | 9 months
Problem Areas In Diabetes-Korean questionnaire at 9 months | 9 months
Patient Satisfaction Questionnaire-Korean at 9 months | 9 months
Cost-effectiveness of pharmaceutical care at 9 months | 9 months